CLINICAL TRIAL: NCT04390698
Title: Opioid Free Anesthesia in Breast Cancer Surgery: a Prospective Randomized Study
Brief Title: Opioid Free Anesthesia in Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Chief of the Anesthesiology Department, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OFA
Record Dates: First submitted 2020-05-08; First posted 2020-05-15 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Opioid Free Anesthesia
MeSH Terms: interventions — Nerve Block; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nerve block+opioid-free general anesthesia (Experimental): Paravertebral block with an ultrasound-guided technique; opioid-free general anesthesia
  Interventions: Procedure: paravertebral block; Drug: opioid free anesthesia
- sham bock+opioid general anesthesia (Sham Comparator): Sham block by local infiltration at the same site of paravertebral block; opioid based general aneshesia
  Interventions: Procedure: sham block; Procedure: opioid general anesthesia

INTERVENTIONS:
Procedure: paravertebral block — Paravertebral block will be performed at T2,T4 level on the surgical side using out-of-plane approach under ultrasound-guided, with 0.4% ropivacaine 20ml at each injection site.
  Other Names: nerve block
  Arms: nerve block+opioid-free general anesthesia
Drug: opioid free anesthesia — propofol, lidocine and muscle relaxant will be used for induction, after laryngeal mask airway insertion, general anesthesia will be maintained.
  Other Names: opioid free
  Arms: nerve block+opioid-free general anesthesia
Procedure: sham block — Local infiltration at the same site of paravertebral block will be performed, with 1% lidocaine 3ml on each injection site.
  Other Names: local infiltration
  Arms: sham bock+opioid general anesthesia
Procedure: opioid general anesthesia — propofol, sufentanil and muscle relaxant will be used for induction, after laryngeal mask airway insertion, general anesthesia will be maintained .
  Other Names: traditional general aneshesia
  Arms: sham bock+opioid general anesthesia

SUMMARY:
A comparison of incidences of postoperative nausea and vomiting (PONV) , postoperative pain severity and recovery parameters in breast cancer patients receiving opioid or opioid-free general anesthesia.

DETAILED DESCRIPTION:
Breast cancer is one of the most common oncologic diagnosis in women. Surgery is traditionally performed under general anesthesia with opioid-based analgesia. It is associated with higher incidences of PONV, more severe acute postoperative pain and increased incidences of chronic pain. The possibility of higher risk of metastasis has also been reported.

The purpose of our study is to compare the opioid-free general anesthesia with the opioid-based general anesthesia with respect to the quality of recovery, postoperative pain and cancer recurrence and metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. first diagnosis of histologically confirmed primary breast cancer without known extension beyond the breast and axillary nodes;
2. ASA physical statue I-II;

Exclusion Criteria:

1. chronic pain and opioid administration history;
2. allergy to local anesthetics or NSAIDs;
3. coagulation disorders;
4. local infection at regional block site;
5. unable to comply to study protocol schedule for logistic or other reasons;
6. refusal to participate to the study；
7. breast reconstruction with implants or latissimus dorsi flap

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
quality of recovery | 24 hours after surgery
  15-item 15-item 15-item quality of recovery questionnaire

SECONDARY OUTCOMES:
health related quality of life | up to 3 months after surgery
  evaluated using EuroQol 5 dimensions questionnaire
postoperative pain | up to 3 months after surgery
  Numeric Rating Scale pain scores, pain questionnaires
cancer recurrence and metastasis | up to 12 months after surgery
  diagnosed by breast cancer specialist

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, MD,PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tripathy S, Rath S, Agrawal S, Rao PB, Panda A, Mishra TS, Nayak S. Opioid-free anesthesia for breast cancer surgery: An observational study. J Anaesthesiol Clin Pharmacol. 2018 Jan-Mar;34(1):35-40. doi: 10.4103/joacp.JOACP_143_17. PMID 29643620
- [Derived] Zhang Q, Wu Y, An H, Feng Y. Postoperative recovery after breast cancer surgery: A randomised controlled trial of opioid-based versus opioid-free anaesthesia with thoracic paravertebral block. Eur J Anaesthesiol. 2023 Aug 1;40(8):552-559. doi: 10.1097/EJA.0000000000001856. Epub 2023 May 23. PMID 37218631